CLINICAL TRIAL: NCT03579433
Title: Postmarket Study of ORA With VerifEye+ and Barrett Toric Calculator Used for the Implantation of AcrySof Toric
Brief Title: Postmarket Study of an Intraocular Lens Power Selection System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILX369-P001
Record Dates: First submitted 2018-06-26; First posted 2018-07-06 (Actual); Results first posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Cataract
Keywords: IOL; Intraocular lens; Astigmatism; Cataract Surgery
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- ORA with VerifEye+ (Experimental): First surgical eye randomly assigned to Acrysof® IQ Toric IOL and ORA with VerifEye+ or Acrysof® IQ Toric IOL and Barrett Toric Calculator, with the second surgical eye (fellow eye) assigned to the alternative group.
  Interventions: Device: ORA with VerifEye+; Device: Acrysof® IQ Toric IOL
- Barrett Toric Calculator (Active Comparator): First surgical eye randomly assigned to Acrysof® IQ Toric IOL and ORA with VerifEye+ or Acrysof® IQ Toric IOL and Barrett Toric Calculator, with the second surgical eye (fellow eye) assigned to the alternative group.
  Interventions: Other: Alcon Barrett Toric Calculator; Device: Acrysof® IQ Toric IOL

INTERVENTIONS:
Device: ORA with VerifEye+ — Intraoperative device that measures total corneal astigmatism in the aphakic condition and is used for the selection of IOL power. In the pseudophakic condition, ORA provides guidance for the alignment of the toric axis mark.
  Arms: ORA with VerifEye+
Other: Alcon Barrett Toric Calculator — Web-based software application that utilizes an algorithm (Barrett Formula) to estimate the amount of post-operative corneal astigmatism in order to optimize IOL model selection and axis placement, with interoperative axis alignment done manually.
  Arms: Barrett Toric Calculator
Device: Acrysof® IQ Toric IOL — Intraocular lens implanted as a replacement for the cataractous lens during cataract surgery (Model SN6AT3, SN6AT4, Model SN6AT5, Model SN6AT6)

SUMMARY:
The purpose of the study was to evaluate the visual acuity outcomes when using the Optiwave Refractive Analysis (ORA) with VerifEye+ and Barrett Toric Calculator for calculating intraocular lens (IOL) power and axis in subjects requiring cataract surgery and implanted with a toric IOL in both eyes.

DETAILED DESCRIPTION:
Surgery was done on each eye on different days, 7 to 14 days apart. Subjects were seen for a total of 10 visits with a follow-up duration of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Planned cataract surgery with IOL implantation
* Able to comprehend and sign the informed consent form
* Preoperative astigmatism of 0.75 to 3.00 Diopter
* Willing and able to complete all required postoperative visits
* Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* Unclear intraocular media other than cataract
* Pregnant or lactating
* Presence or history of any condition or finding that makes the subject unsuitable as a candidate for cataract surgery or study participation or may confound the outcome of the study, in the opinion of the Investigator.
* Other protocol-defined exclusion criteria may apply

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Operations Lead, Surgical, Study Director — Alcon Research, LLC
Locations (9):
- United States (9):
  - Alcon Investigative Site, Mt. Dora, Florida
  - Alcon Investigative Site, Panama City, Florida
  - Alcon Investigative Site, Poughkeepsie, New York
  - Alcon Investigative Site, Kingston, Pennsylvania
  - Alcon Investigative Site, Florence, South Carolina
  - Alcon Investigative Site, Mt. Pleasant, South Carolina
  - Alcon Investigative Site, Sioux Falls, South Dakota
  - Alcon Investigative Site, Nashville, Tennessee
  - Alcon Investigative Site, Nacogdoches, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 124 subjects enrolled, 12 subjects were discontinued prior to randomization, and 8 subjects were randomized, but not treated in either eye. This reporting group includes all subjects with attempted implantation of an intraocular lens (IOL) in one or both eyes.
Groups:
- All Participants: First surgical eye randomly assigned to Acrysof® IQ Toric IOL and Optiwave Refractive Analysis with VerifEye+ (ORA With VerifEye+) or Acrysof® IQ Toric IOL and Barrett Toric Calculator (Barrett Toric Calculator), with the second surgical eye (fellow eye) assigned to the alternative group.
Period: Overall Study
Arm/Group | All Participants
Started | 104
ORA With VerifEye+ (Successful implantation) | 96
Barrett Calculator (Successful implantation) | 102
Completed | 98
Not Completed | 6

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Groups:
- Overall: First surgical eye randomly assigned to Acrysof® IQ Toric (IOL) and Optiwave Refractive Analysis (ORA) with VerifEye+ or Acrysof® IQ Toric IOL and Barrett Toric Calculator, with the second surgical eye (fellow eye) assigned to the alternative group.
Arm/Group | Overall
Number analyzed (Participants) | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.0 (8.73)
Age, Customized [Count of Participants; unit: Participants]
  Less than 65 years old | 28
  65 years old or older | 76
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 102
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 96
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 104

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eyes With Best Corrected Distance Visual Acuity (BCDVA) of 20/20 or Better at Month 6
Description: Visual acuity (VA) was tested monocularly (each eye separately) using the correction obtained from the manifest refraction and 100% contrast electronic Early Treatment Diabetic Retinopathy Study (ETDRS) charts at a distance of 4 meters (m) from the eye. 20/20 represents normal distance eyesight. No hypothesis testing of the primary endpoint was specified.
Time Frame: Month 6
Population: The Per Protocol Analysis Set (PPS) includes all eyes with successful IOL implantation, T3-T6 and recommended by ORA and with no major protocol deviations and data at visit.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Groups:
- ORA With VerifEye+: Acrysof® IQ Toric IOL and ORA with VerifEye+
- Barrett Toric Calculator: Acrysof® IQ Toric IOL and Barrett Toric Calculator
Arm/Group | ORA With VerifEye+ | Barrett Toric Calculator
Number analyzed (Participants) | 85 | 95
Number analyzed (eyes) | 85 | 95
percentage of eyes | 87.1 | 87.4

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of attempted implantation with any IOL through study completion, an average of 120-180 days.
Description: Adverse events were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator as outlined in the study protocol. "At Risk" population for ocular adverse events is included with unit of "eyes."
Groups:
- Pretreatment: All subjects prior to with attempted implantation with any IOL (successful or aborted after contact with the eye)
- ORA With VerifEye+ Study Eye: All eyes with attempted implantation (successful or aborted after contact with the eye) of Acrysof® IQ Toric IOL and ORA with VerifEye+
- Barrett Toric Calculator Study Eye: All eyes with attempted implantation (successful or aborted after contact with the eye) of Acrysof® IQ Toric IOL and Barrett Toric Calculator
- Overall Systemic: All subjects with attempted implantation with any IOL (successful or aborted after contact with the eye)
Arm/Group | Pretreatment | ORA With VerifEye+ Study Eye | Barrett Toric Calculator Study Eye | Overall Systemic
All-Cause Mortality (participants affected / at risk) | 0/104 | 0/96 | 0/102 | 0/104
Serious Adverse Events (participants affected / at risk) | 0/104 | 2/96 | 2/102 | 1/104
Other Adverse Events (participants affected / at risk) | 0/104 | 10/96 | 7/102 | 0/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pretreatment (N=104) | ORA With VerifEye+ Study Eye (N=96) | Barrett Toric Calculator Study Eye (N=102) | Overall Systemic (N=104)
Metamorphopsia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Assessed as not related to the Barrett Toric Calculator
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Assessed as not related to the ORA With VerifEye
Retinal tear (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Assessed as not related to the ORA With VerifEye
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye laser surgery (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — Assessed as not related to the ORA With VerifEye
Intraocular lens implant (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Assessed as not related to the Barrett Toric Calculator
Intraocular lens repositioning (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (2) | 0 (0) — Assessed as not related to the Barrett Toric Calculator
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pretreatment (N=104) | ORA With VerifEye+ Study Eye (N=96) | Barrett Toric Calculator Study Eye (N=102) | Overall Systemic (N=104)
Posterior capsule opacification (Eye disorders) | 0 (0) | 5 (5) | 3 (3) | 0 (0) — Assessed as not related to the ORA with VerifEye or Barrett Toric Calculator
Intraocular pressure increased (Investigations) | 0 (0) | 7 (7) | 4 (4) | 0 (0) — Assessed as not related to the ORA with VerifEye or Barrett Toric Calculator

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/33/NCT03579433/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-22): https://cdn.clinicaltrials.gov/large-docs/33/NCT03579433/SAP_001.pdf